CLINICAL TRIAL: NCT03623776
Title: A Multicenter Phase II Trial of Neoadjuvant JS001, or JS001 in Combination With Chemotherapy in Resectable NSCLC.
Brief Title: Neoadjuvant JS001, or JS001 in Combination With Pemetrexed and Carboplatin in Resectable NSCLC.
Acronym: NAJSCR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients enrolled.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Si-Yu Wang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO1038
Record Dates: First submitted 2018-07-30; First posted 2018-08-09 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Efficacy and Safety
Keywords: Non-Small Cell Lung Cancer; Neoadjuvant; Programmed Death-1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — toripalimab; Pemetrexed; Carboplatin; Thoracic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS001 alone (Experimental): Subjects receive JS001 240 mg i.v. infusion on Day 1 of each 21-day cycle for 3 cycles.
  Interventions: Drug: JS001; Procedure: Thoracic Surgery
- JS001+chemotherapy (Experimental): Subjects receive JS001 240 mg, pemetrexed of 500 mg/m^2 and carboplatin at the AUC of 5 administered as IV infusion on Day 1 of each 21-day cycle for 3 cycles.
  Interventions: Drug: JS001; Drug: Pemetrexed; Drug: Carboplatin; Procedure: Thoracic Surgery

INTERVENTIONS:
Drug: JS001 — JS001 was given 240 mg i.v. infusion on Day 1 of each 21-day cycle for 3 cycles.
  Other Names: Toripalimab
Drug: Pemetrexed — Subjects receive pemetrexed of 500 mg/m^2 administered as IV infusion on Day 1 of each 21-day cycle for 3 cycles.
  Other Names: Pemetrexed Disodium
  Arms: JS001+chemotherapy
Drug: Carboplatin — Subjects receive carboplatin at the AUC of 5 administered as IV infusion on Day 1 of each 21-day cycle for 3 cycles.
  Other Names: CBP
  Arms: JS001+chemotherapy
Procedure: Thoracic Surgery — Surgery will be performed at least 21 days after the last dose of neoadjuvant therapy.

SUMMARY:
JS001 (Toripalimab) is a recombinant humanized anti-PD-1 monoclonal antibody, which selectively interferes with the combination of PD-1 with its ligands, PD-L1 and PD-L2. The purpose of this study is to studying neoadjuvant JS001, or JS001 in combination with pemetrexed and carboplatin to see how well it works in treating patients with resectable NSCLC.

DETAILED DESCRIPTION:
Surgery in combination with preoperative or postoperative chemotherapy is the recommended therapeutic approach for patients with resectable non-small cell lung cancer (NSCLC). However, the prognosis of early-stage NSCLC remains to be improved, with 5-year survival rates ranging from 50% for stage IA to 20% for stage IIIA. Antibodies that block the PD-1 protein have provided a major treatment advance in patients with cancer. JS001 (Toripalimab) is a recombinant humanized anti-PD-1 monoclonal antibody, which has shown its efficacy in the treatment of a variety of malignancies. This study is to studying neoadjuvant JS001, or JS001 in combination with chemotherapy to see how well it works in treating patients with resectable NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Target population is high risk NSCLC with resection option for potential cure, as assessed by a faculty surgeon at SYSUCC. This may include clinical stage IB (≥4cm), II and IIIA. Subjects with N3 nodal involvement are not included.
* Subjects should not have a previously detected sensitizing EGFR mutation or ALK fusion oncogene.
* Written informed consent provided.
* Male and female patients aged ≥18 years, < 75 years.
* Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
* Blood and specimens before and after treatment must be provided
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Life expectancy ≥12 weeks.
* Adequate hematological function: Absolute neutrophil count (ANC) ≥2.0 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level).
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN), Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN in subjects without liver metastases; ≤ 5 x ULN in subjects with liver metastases.
* Adequate renal function: Serum creatinine ≤ 1.25 x ULN, or ≥ 60 ml/min.
* Female subjects should not be pregnant or breast-feeding.

Exclusion Criteria:

* Known severe hypersensitivity to JS001 or any of the excipients of this product.
* Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody (including any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Prior chemotherapy or radiotherapy.
* Subjects with active, known or suspected autoimmune disease. Subjects in conditions not expected to recur in the absence of an external trigger, or not requiring systemic treatment are permitted to enroll.
* Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first administration of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Inability to comply with protocol or study procedures.
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* A serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease.
* History of another malignancy in the last 5 years with the exception of the following: other malignancies cured by surgery alone and having a continuous disease-free interval of 5 years are permitted. Cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix are permitted.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
* Patient who has active serious infection (e.g. pyrexia of or 38.0℃ over)
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Known history of active Hepatitis B or C.
* Women who are pregnant or nursing.
* Evidence of any other disease, neurological or metabolic dysfunction, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that contraindicated the use of an investigational drug or puts the subject at high risk for treatment-related complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
3-year Disease Free Survival | 3 years after the last patient is registered
  Disease-free survival was assessed from registration to disease recurrence or death as a result of any cause.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events (AEs) | 2 years after the last patient is registered
  Adverse Events were monitored according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0.
Number of participants with perioperative complications | 2 years
  Perioperative complications will be recorded
3-year Overall survival | 3 years after the last patient is registered
  Overall survival was assessed from registration to death as a result of any cause.
Pathologic Response | 3 months
  To assess pathologic response to neoadjuvant JS001, or JS001 in combination with chemotherapy in resected tumor and lymph nodes. Major pathologic response was defined as <10% residual viable tumor cells in the resection specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Si-Yu Wang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes